CLINICAL TRIAL: NCT03936192
Title: Parallel-group Active Comparator, Double-blind, Randomized, Phase III Study to Assess Safety, Efficacy of Glucosamine Sulfate Plus Meloxicam vs Glucosamine Sulfate Plus Chondroitin Sulfate Primary Symptomatic Knee Osteoarthritis Treatment
Brief Title: A Parallel-group Active Comparator, Double-blind, Multicenter, Randomized, Double-blind, Phase III Clinical Study
Acronym: SAVE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EF 156
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucosamine; Meloxicam; Chondroitin Sulfates

STUDY DESIGN:
Intervention Model Description: glucosamine sulphate 1500mg + meloxicam 15mg, produced by Eurofarma Laboratories S.A., administered once a day for 12 weeks.
  Glucosamine sulfate 1500mg + Chondroitin sulfate 1200mg, produced by Zodiac Pharmaceutical Products S.A. (Condroflex®), given once daily for 12 weeks.
  Placebo administered once daily for 12 weeks.
Who Masked: Participant, Investigator
Masking Description: Participant and Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- glucosamine sulfate 1500mg and meloxicam 15mg (Eurofarma) (Experimental): glucosamine sulfate 1500mg plus meloxicam 15mg combination, manufactured by Eurofarma Laboratories S.A., administered once a day for 12 weeks.
  Interventions: Drug: glucosamine sulphate 1500mg and meloxicam 15mg
- Glucosamine sulfate 1500mg and chondroitin sulfate 1200mg (Active Comparator): Glucosamine sulfate 1500mg plus Chondroitin Sulfate 1200mg, manufactured by Zodiac Pharmaceutical Products S.A. (Condroflex®), given once daily for 12 weeks.
  Interventions: Drug: Glucosamine sulfate 1500mg and chondroitin sulfate 1200mg
- Placebo (Placebo Comparator): Placebo administered once daily for 12 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: glucosamine sulphate 1500mg and meloxicam 15mg — glucosamine sulphate 1500mg plus meloxicam 15mg, manufactured by Eurofarma Laboratories S.A., administered once a day for 12 weeks.
  Other Names: glucosamine sulfate 1500mg and meloxicam 15mg (Eurofarma)
  Arms: glucosamine sulfate 1500mg and meloxicam 15mg (Eurofarma)
Drug: Glucosamine sulfate 1500mg and chondroitin sulfate 1200mg — Glucosamine sulfate 1500mg and chondroitin sulfate 1200mg, manufactured by Zodiac Pharmaceutical Products S.A. (Condroflex®)
  Other Names: glucosamine sulfate 1500mg and chondroitin sulfate 1200mg (Eurofarma)
  Arms: Glucosamine sulfate 1500mg and chondroitin sulfate 1200mg
Drug: Placebos — Placebo administered once daily for 12 weeks.
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, parallel-group, placebo-controlled, and active-drug, 12-week, multicenter clinical study. Participants will be randomized 2: 2: 1 to receive the combination of glucosamine sulfate + meloxicam (experimental group), combination of glucosamine sulfate + chondroitin sulfate (active control group) or placebo.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, parallel-group, placebo-controlled, and active-drug, 12-week treatment period, phase 3 comparative clinical study. Participants will be randomized 2:2:1 to receive the combination of glucosamine sulfate + meloxicam (experimental group), combination of glucosamine sulfate + chondroitin sulfate (active control group) or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 40 to 75 years (both inclusive).
2. Clinical and radiological diagnosis of primary (idiopathic) knee osteoarthritis according to the American College of Rheumatology (ACR) criteria.
3. Radiological classification of Kellgren and Lawrence of grades 2 or 3 on X-ray of the target knee.
4. Presence of painful symptoms in the target knee in the last 3 months due to osteoarthritis.
5. Visual analogue scale for evaluation of knee osteoarthritis pain by the research participant ≥ 40 mm at the screening visit.
6. Mean score ≥ 40mm on the "pain" subscale (0 to 100mm) on the target knee of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire at the randomization visit.
7. ACR functional class from I to III.
8. Signature of the Informed Consent Form before performing any study procedure.

Exclusion Criteria:

1. Diagnosis of septic arthritis, inflammatory arthritis (such as rheumatoid arthritis), gout, pseudogout, Paget's disease, dysplasias or congenital articular anomalies.
2. Severe joint misalignment in the target knee, defined by the researcher.
3. History of severe trauma or surgery (including arthroscopy) in the target knee within 6 months prior to the study selection visit.
4. Symptomatic osteoarthritis of the ipsilateral hip.
5. Use of non-steroidal anti-inflammatory, dipyrone, opioid or narcotic analgesics, collagen and herbal remedies for osteoarthritis from the screening visit, or a washout period for such drugs less than those defined by the protocol, prior to the visit randomization. The use of antidepressants and pain modulating medicinal products should not be started from the screening visit, but they should be kept stable during the study if they are already being used prior to the screening visit.
6. Oral, intravenous or intramuscular corticosteroid therapy within 30 days prior to study visit visit.
7. Intra-articular injection of corticosteroids, hyaluronic acid and / or platelet-rich plasma at the target knee within 6 months prior to the study selection visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
To assess whether the efficacy of glucosamine + meloxicam sulfate treatment is superior to the efficacy of treatment with glucosamine sulfate + chondroitin sulfate in improving pain in subjects with symptomatic primary knee OA treated for 4 weeks. | 4 weeks
  Absolute variation of the "pain" subscale score of the WOMAC questionnaire (0 to 100mm) 4 weeks (V2) after starting treatment in relation to the basal score (VR);

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.